CLINICAL TRIAL: NCT05433545
Title: Adherence to Physiotherapy Scoliosis Specific Exercises in Adolescents With Spine Deformity: Development of a New Questionnaire
Status: Recruiting | Type: Observational
Sponsor: Istituto Scientifico Italiano Colonna Vertebrale (Other)
Responsible Party: Sponsor
Other Study IDs: AdePSSE
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Adherence, Treatment; Spinal Deformity
MeSH Terms: conditions — Treatment Adherence and Compliance | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adherence to specific physiotherapy exercises
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Adolescents with spinal deformity will be asked to fill out a new questionnaire measuring the quality and quantity of adherence to specific physiotherapy exercises performed at home. Patients will be recruited at an outpatient service dedicated to the treatment of vertebral deformities during the monthly sessions with the physiotherapist

SUMMARY:
This study aims to develop a new instrument capable of providing an efficient measure of the quality and quantity of adherence to Physiotherapy Scoliosis Specific Exercises performed at home by growing patients with spinal deformity undergoing conservative treatment at a specialized institution. The development of a questionnaire in a Rasch environment and specifically developed for this population will ensure greater sensitivity and specificity of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* aged between 10 and 18 years
* adolescent idiopathic scoliosis of 10 ° Cobb or more
* Scheuermann's kyphosis or idiopathic hyperkyphosis
* prescription of specific exercises

Exclusion Criteria:

* positive neurological evaluation

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents with spinal deformity treated with Physiotherapy Scoliosis Specific Exercises
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to Physiotherapy Scoliosis Specific Exercises | through study completion, an average of 1 year
  New questionnaire developped to assess quality and quantity of adherence to specific physiotherapy exercises performed at home patients with spinal deformity treated conservatively

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Vanossi, PT, Principal Investigator — Istituto Scientifico Italiano Colonna Vertebrale
Locations (1):
- ISICO, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: Yes
The raw data will be shared on a repositiry